CLINICAL TRIAL: NCT03339336
Title: A Phase 2 Placebo-Controlled, Double-Blind, Enriched Enrollment Randomized Withdrawal Study to Evaluate the Efficacy and Safety of BIIB074 (Vixotrigine) in Treating Pain Experienced by Subjects With Confirmed Small Fiber Neuropathy That is Idiopathic or Associated With Diabetes Mellitus
Brief Title: Efficacy and Safety Study of BIIB074 in Participants With Small Fiber Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to close study early; not due to safety concerns
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 802NP206; 2017-000991-27 (EudraCT Number)
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Small Fiber Neuropathy; Diabetes Mellitus
MeSH Terms: conditions — Small Fiber Neuropathy; Diabetes Mellitus | interventions — vixotrigine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BIIB074 350 mg (Experimental): Taper Period (if applicable) from neuropathic pain medication, followed by a washout period, then BIIB074 350 mg tablets orally twice daily (BID) Open-Label Run-In Period, then BIIB074 350 mg tablets orally BID Double-Blind Treatment Period.
  Interventions: Drug: BIIB074
- BIIB074 200 mg (Experimental): Taper Period (if applicable) from neuropathic pain medication, followed by a washout period, then BIIB074 350 mg tablets orally twice daily (BID) Open-Label Run-In Period, then BIIB074 200 mg tablets orally BID Double-Blind Treatment Period.
  Interventions: Drug: BIIB074
- Placebo (Placebo Comparator): Taper Period (if applicable) from neuropathic pain medication, followed by a washout period, then BIIB074 350 mg tablets orally twice daily (BID) Open-Label Run-In Period, then BIIB074 placebo-matching tablets orally BID Double-Blind Treatment Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB074 — Administered as specified in the treatment arm.
  Arms: BIIB074 200 mg; BIIB074 350 mg
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of BIIB074 in treating pain experienced by participants with confirmed small fiber neuropathy (SFN) that is idiopathic or associated with diabetes mellitus. A secondary endpoint that relates to the primary objective is the change from Randomization to Week 12 of the double-blind period in mean average daily pain score.

The secondary objectives of this study are to evaluate the effect on worst pain, neuropathic pain quality, sleep interference due to pain, patient global impression, use of rescue medication, and SFN symptoms in participants treated with BIIB074; to investigate the safety and tolerability of BIIB074 in participants with SFN; and to characterize the pharmacokinetics (PK) of BIIB074 in participants with SFN.

ELIGIBILITY:
Key Inclusion Criteria:

1. This study will be conducted in subjects who have had a diagnosis of at least probable SFN, length-dependent distribution, for 6 months and ≤10 years prior to screening, defined as a history of the symptoms and clinical signs based on discussions at the ACTTION CONCEPPT meeting on diagnosis of SFN, Washington, DC March 2018, and confirmed by intraepidermal nerve fiber density (IENFD) values, and weekly mean average daily pain (ADP) score of ≥5 and ≤9 on an 11-point Pain Intensity Numeric Rating Scale (PI-NRS) over the last 7 days of prior to the Screening visit.
2. In addition to these criteria, subjects with diabetes will be required to have HbA1c ≤11%, treated with oral hypoglycemics and/or subcutaneous insulin or diet, no evidence of ulcers, advanced retinopathy (defined as greater than State 3 [moderate non-proliferative diabetic retinopathy]) (DCCT/EDIC Research Group 2017), severe nephropathy, or clinically significant obstructive atherosclerotic disease or current class IV heart failure to be eligible for the study.

Key Exclusion Criteria:

1. Previous exposure to BIIB074 (formerly known as CNV1014802 or GSK1014802).
2. Use of capsaicin patch within 3 months prior to Screening.
3. Unable or unwilling to discontinue concomitant medications for SFN pain prior to Day 1.
4. Unable or unwilling to comply with the prohibited concomitant medication restrictions, including but not limited to UDP-glucuronosyltransferase (UGT) inducers and inhibitors, monoamine oxidase inhibitors (MAOIs), and Nav blockers.
5. Use of over-the-counter medications, vitamin and mineral supplements, herbal remedies (including St. John's wort), dietary supplements, or foods (including grapefruit juice) that affect and UGTs.
6. Unable or unwilling to discontinue medications that are P-glycoprotein substrates with a narrow therapeutic index, including but not limited to digoxin.
7. History of hemophilia or Von Willebrand's disease, or use of anticoagulants that may result in bleeding risk during the skin biopsy.
8. Any contraindication, as determined by the Investigator, to performing a skin biopsy for intraepidermal nerve fiber analysis.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Weekly Mean Average Daily Pain (ADP) Score | Baseline and Week 12 of the Double-Blind Period
  Participants will rate their ADP using an 11-point Numerical Rating Scale (NRS) (0=no pain and 10=worst possible pain) and record their score in an electronic diary (eDiary). Weekly mean ADP scores for Baseline (the 5 days prior to the first dose of study treatment in the open-label run-in period) and Week 12 (the 7 days prior to the visit at the end of Week 12) will be derived from the ADP scores and calculated as the mean of the daily scores over the last 7 days.
Change from Randomization in Weekly Mean ADP Score | Randomization and Week 12 of the Double-Blind Period
  Participants will rate their ADP using an 11-point NRS (0=no pain and 10=worst possible pain) and record their score in an eDiary. Weekly mean ADP scores for Randomization (the 7 days prior to the first dose of study treatment in the double-blind period) and Week 12 (the 7 days prior to the visit at the end of Week 12) will be derived from the ADP scores and calculated as the mean of the daily scores over the last 7 days.

SECONDARY OUTCOMES:
Change from Baseline in Weekly Mean Worst Daily Pain (WDP) Score | Baseline and Week 12 of the Double-Blind Period
  Participants will rate their WDP using an 11-point NRS (0=no pain and 10=worst possible pain) and record their score in an eDiary. Weekly mean WDP scores for Baseline (the 5 days prior to the first dose of study treatment in the open-label run-in period) and Week 12 (the 7 days prior to the visit at the end of Week 12) will be derived from the WDP scores and calculated as the mean of the daily scores over the last 7 days.
Change from Baseline in Weekly Mean Sleep Interference Numerical Rating Scale (S-NRS) | Baseline and Week 12 of the Double-Blind Period
  Participants will rate their S-NRS using an 11-point NRS (0=pain does not interfere with sleep and 10= pain completely interferes with sleep) and record their score in an eDiary. Weekly mean S-NRS scores for Baseline (the 5 days prior to the first dose of study treatment in the open-label run-in period) and Week 12 (the 7 days prior to the visit at the end of Week 12) will be derived from the daily S-NRS scores and calculated as the mean of the daily scores over the last 7 days.
Change from Baseline in Neuropathic Pain Symptom Inventory (NPSI) Total Score and Sum Score | Baseline and Week 12 of Double-Blind Period
  Participant will use the NPSI questionnaire to rate different symptoms of neuropathic pain. The NPSI includes ten items related to different pain descriptors (e.g. burning and pressure) that are rated on an 11-point NRS (0=no symptoms to 10=worst symptoms imaginable). A score in each dimension and also a total score (from 0-100) is generated using data from the questionnaire.
Proportion of Participants with at least a 2-point Reduction from Baseline in Weekly Mean ADP | Baseline and Week 12 of the Double-Blind Period
  Participants will rate their ADP using an 11-point NRS (0=no pain and 10=worst possible pain) and record their score in an electronic diary (eDiary). Weekly mean ADP scores for Baseline (the 5 days prior to the first dose of study treatment in the open-label run-in period) and Week 12 (the 7 days prior to the visit at the end of Week 12) will be derived from the ADP scores and calculated as the mean of the daily scores over the last 7 days.
Proportion of Participants with at least a 30% Reduction from Baseline in Weekly Mean ADP | Baseline and Week 12 of Double-Blind Period
  Participants will rate their ADP using an 11-point NRS) (0=no pain and 10=worst possible pain) and record their score in an electronic diary (eDiary). Weekly mean ADP scores for Baseline (the 5 days prior to the first dose of study treatment in the open-label run-in period) and Week 12 (the 7 days prior to the visit at the end of Week 12) will be derived from the ADP scores and calculated as the mean of the daily scores over the last 7 days.
Mean Weekly Amount of Rescue Medication | Weekly from Baseline to Week 12 of the Double-Blind Period
  Use of rescue medication (paracetamol/acetaminophen) will be monitored and dosage will be recorded on a daily basis by the participant using an electronic Diary (eDiary). Mean weekly amount of rescue medication used for neuropathic pain during the double-blind period.
Patient Global Impression of Change (PGIC) | Week 12 of the Double-Blind Period
  PGIC is a 7-point self-administered scale that depicts changes in a participant's overall status. Participants will rate their change as "1=very much improved," "2=much improved," "3=minimally improved," "4=no change," "5=minimally worse," "6=much worse," or "7=very much worse."
Change from Baseline in Brief Pain Inventory-Short Form (BPI-SF) Interference Score | Baseline and Week 12 of the Double-Blind Period
  The BPI-SF is a 7-item self-administered questionnaire that measures how much pain has interfered with daily functioning. Participants will rate the level of pain interference on daily functioning on an 11-point NRS where 0=does not interfere and 10=completely interferes.
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) During Double-Blind Period | Week 5 to Week 17
  AEs: any sign, symptom, or diagnosis/disease that is unfavorable or unintended, that is new, or if pre-existing, worsens in participants administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. SAEs: an event that results in death; an event that, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event); an outcome that results in a congenital anomaly/birth defect diagnosed in a child of a participant; an event that requires or prolongs inpatient hospitalization; an event that results in persistent or significant disability/incapacity. Any other medically important event that, in the opinion of the investigator, may jeopardize the participant or may require intervention to prevent one of the other outcomes listed in the definition above.
Area Under the Concentration-time Curve at Steady State | Week 1, 3, 5, 9, 13 and 17 prior to dosing and 1 to 2 hours after dosing, and at Day 123 (Follow-up clinic visit)
Maximum Observed Concentration (Cmax) at Steady State | Week 1, 3, 5, 9, 13 and 17 prior to dosing and 1 to 2 hours after dosing, and at Day 123 (Follow-up clinic visit)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (97):
- Bulgaria (4):
  - Research Site, Byala
  - UMHAT 'Dr Georgi Stranski' EAD, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (7):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Toronto General Hospital, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Recherche Médicale St-Jérôme Inc., Saint-Jérôme, Quebec
  - Research Site, Kingston
  - Research Site, Winnipeg
- Czechia (6):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice u sv. Anny v Brne, Brno
  - Research Site, Hradec Králové
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Nemocnice Pardubickeho kraje a.s. Pardubicka nemocnice, Pardubice
  - Fakultni nemocnice v Motole, Prague
- Denmark (4):
  - Research Site, Aarhus
  - Research Site, Copenhagen
  - Research Site, Herlev
  - OUH, Odense
- France (12):
  - Research Site, Brest, Finistere
  - Hopital Salengro - CHRU de Lille, Lille, Nord
  - CHU Saint Etienne - Hôpital Nord, Saint Priest En Jarez, Pays de la Loire Region
  - CHU Clermond Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand, Puy De Dome
  - Research Site, Vénissieux, Rhone
  - Hôpital Ambroise Paré - Boulogne-Billancourt, Boulogne-Billancourt
  - Research Site, Corbeil-Essonnes
  - Hopital Henri Mondor, Créteil
  - Research Site, Le Creusot
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU Nice - Hôpital de l'Archet 1, Nice
  - Hopital Lariboisiere, Paris
- Germany (14):
  - Clinical Research, Böblingen, Baden-Wurttemberg
  - Research Site, Aschaffenburg, Bavaria
  - Research Site, Künzing, Bavaria
  - Clinical Research, Westerstede, Lower Saxony
  - Clinical Research, Münster, Nord Rhein Westfalen
  - Gemeinschaftspraxis Diabeteszentrum Dortmund Dr.med. Klaus Busch, Dortmund, North Rhine-Westphalia
  - Hausarzt- und Diabetologische Schwerpunktpraxis, Lage, Saxony-Anhalt
  - Zentrum fur Klinische Forschung, Bad Homburg
  - Gemeinschaftspraxis für Neurologie, Berlin
  - Research Site, Essen
  - Diabetologische Schwerpunktpraxis Harburg, Hamburg
  - Research Site, Mainz
  - DKD Helios Klinik Wiesbaden, Wiesbaden
  - Research Site, Würzburg
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Pátrai
  - AHEPA General Hospital of Thessaloniki, Thessaloniki
- Hungary (7):
  - Research Site, Baja
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaz, Békéscsaba
  - UNO Medical Trials Kft., Budapest
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
- Italy (6):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Research Site, Genova
  - Research Site, Milan
  - Azienda Ospedaliero Univeraitaria Pisana, Pisa
  - Università Campus Bio-Medico di Roma, Roma
  - Research Site, Telese Terme
- Netherlands (2):
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Maastricht UMC+, Maastricht
- Poland (8):
  - Research Site, Bydgoszcz
  - Research Site, Chorzów
  - PRATIA MCM Kraków, Krakow
  - Research Site, Lublin
  - Research Site, Oświęcim
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - Research Site, Warsaw
  - Regionalna Poradnia Diabetologiczna Zytkiewicz-Jaruga,Stasinska, Wroclaw
- Spain (8):
  - Research Site, A Coruña
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitari de Bellvitge, Barcelona
  - Research Site, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Research Site, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitari i Politecnic La Fe, Valencia
- Switzerland (4):
  - CHUV - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Ospedale Regionale di Lugano, Lugano
  - Kantonspital St. Gallen, Sankt Gallen
  - Research Site, Zurich
- United Kingdom (11):
  - Royal Hallamshire Hospital, Sheffield, South Yorkshire
  - Clinical Reseach, Bath
  - Research Site, Ipswich
  - Research Site, Liverpool
  - Guy's Hospital, London
  - King's College Hospital, London
  - St Pancras Clinical Research, London
  - The Royal London Hospital, London
  - Research Site, Manchester
  - John Radcliffe Hospital, Oxford
  - Research Site, Swansea

REFERENCES:
- [Derived] Faber CG, Attal N, Lauria G, Dworkin RH, Freeman R, Dawson KT, Finnigan H, Hajihosseini A, Naik H, Serenko M, Morris CJ, Kotecha M. Efficacy and safety of vixotrigine in idiopathic or diabetes-associated painful small fibre neuropathy (CONVEY): a phase 2 placebo-controlled enriched-enrolment randomised withdrawal study. EClinicalMedicine. 2023 Apr 27;59:101971. doi: 10.1016/j.eclinm.2023.101971. eCollection 2023 May. PMID 37152360